CLINICAL TRIAL: NCT06170216
Title: A Single-center, Non-interventionary Clinical Study Evaluating the Efficacy and Safety of Different Immunochemotherapies in Small B-cell Non-Hodgkin Lymphoma (iNHL)
Brief Title: Different Immunochemotherapies in Small B-cell Non-Hodgkin Lymphoma (iNHL)
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yizhen Liu, Clinical Professor, Fudan University
Other Study IDs: iNHL-01
Record Dates: First submitted 2023-11-29; First posted 2023-12-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iNHL: Different immunochemotherapies in small B-cell non-Hodgkin lymphoma
  Interventions: Drug: immunochemotherapies

INTERVENTIONS:
Drug: immunochemotherapies — Observing different immunochemotherapies in small B-cell non-Hodgkin lymphoma (iNHL), which are chosen by investigators, such as RCHOP, BR, RCVP, etc.

SUMMARY:
Describe the application status of different immunochemotherapies in small B-cell non-Hodgkin lymphoma (iNHL), observe the therapeutic efficacy and safety of the treatment modalities.

DETAILED DESCRIPTION:
Evaluated the efficacy and safety of different immunochemotherapies in small B-cell non-Hodgkin lymphoma (iNHL)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Initial or first recurrent iNHL confirmed by histopathology, including FL (1-3a), MZL, MCL;
* Sign an informed consent form;
* Researchers evaluate patients who can benefit from receiving immunochemotherapy.

Exclusion Criteria:

* There are contraindications to any medication in the treatment plan;
* Pregnant or lactating women or male and female participants of childbearing age did not take contraceptive measures during the trial period and within 30 days after the last medication;
* Researchers believe that patients who are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibale patients who ≥ 18 years old, Initial or first recurrent iNHL, with no contraindications to any medication in the treatment plan are enrolled. They will sign an informed consent form. Pregnant or lactating women were excluded. And patients who may not benefit from receiving immunochemotherapy evaluated by researchers are also excluded.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 6 months
  the ratio of numbers of patients with complete response and partial response to all the participants receiving treatment

SECONDARY OUTCOMES:
2-year progression-free survival (PFS) | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason
2-year event-free survival (EFS) | From date of patients sign informed consent until the date of first documented event, progression or date of death from any cause, whichever came first, assessed up to 2 years
  the period from the date of patients sign informed consent to the observed event for any reason
overall survival | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 2 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time
Hematology and non hematology toxicity | Throughout the treatment period，up to 6 months
  number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided